CLINICAL TRIAL: NCT05778318
Title: Efficacy of Lianhua Qingwen in Treating Patients Infected With the Omicron Variant of the COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Qian Qi, Dr., Qianfoshan Hospital
Other Study IDs: YXLL-KY-2022(095)
Record Dates: First submitted 2023-03-20; First posted 2023-03-21 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients without Lianhua Qingwen treatment.
  Interventions: Other: The group of patients who did not receive Lianhua Qingwen orally
- Observation Group: Patients with Lianhua Qingwen treatment.
  Interventions: Drug: The group of patients who received Lianhua Qingwen orally

INTERVENTIONS:
Drug: The group of patients who received Lianhua Qingwen orally — Lianhua Qingwen Granules: oral. One bag at a time, three times a day. The course of treatment for mild and ordinary cases of novel coronavirus pneumonia is 7-10 days.
  Groups: Observation Group
Other: The group of patients who did not receive Lianhua Qingwen orally — The group of patients who did not receive Lianhua Qingwen orally.
  Groups: Control group

SUMMARY:
A retrospective analysis was conducted on patients infected with the Omicron variant of COVID-19 diagnosed from August 2022 to now. Patients were divided into observation groups and control groups according to whether or not oral Lianhua Qingwen granules were used. Through data analysis and follow-up, the effectiveness of Lianhua Qingwen in treating patients infected with the Omicron variant of COVID-19 was discussed.

ELIGIBILITY:
Inclusion Criteria:

* For patients infected with the Omicron variant, the diagnostic criteria are confirmed cases of COVID-19 and clinical classification according to the diagnostic criteria of Prevention and Control Protocol for COVID-19 (Trial Eighth Edition) issued by the National Health and Construction Commission.
* The clinical symptoms were classified as mild or ordinary.
* They have been vaccinated against the COVID-19.

Exclusion Criteria:

* Patients receiving antiviral or antibiotic drugs
* Severe and critical patients with COVID-19.
* Patients with chronic respiratory diseases, bacterial infections of the respiratory system, and other respiratory diseases affecting the study.
* Patients with serious primary diseases of the heart, brain, lung, liver, kidney, and hematopoietic systems, as well as mental diseases.
* Allergic reaction to Lianhua Qingwen granules.
* Excluded patients treated with the same drug as Lianhua Qingwen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ① For patients infected with the Omicron variant of COVID-19, the diagnostic criteria are confirmed cases of COVID-19 and clinical classification according to the diagnostic criteria of Prevention and Control Protocol for Novel Coronavirus Pneumonia (Trial Eighth Edition) issued by the National Health and Construction Commission; ② The clinical symptoms were classified as mild or ordinary; ③ They have been vaccinated against the COVID-19.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Disappearance rate of symptoms | two weeks
  Disappearance rate of symptoms (fever, fatigue, cough)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, #16766, Jingshi Road, Jinan City, Shandong Province, China, Jinan, Shandong, China